CLINICAL TRIAL: NCT01499316
Title: Investigating the Effects of Hyperoxia on Fractional Flow Reserve in Patients With Moderate Coronary Artery Disease
Brief Title: Investigating the Effects of Hyperoxia on Fractional Flow Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 426/11
Record Dates: First submitted 2011-12-05; First posted 2011-12-26 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flow oxygen (Experimental): 10 minute of 10/L min of inhaled oxygen with reservoir bag.
  Interventions: Procedure: High Flow oxygen
- Room Air (Experimental)
  Interventions: Procedure: Room Air

INTERVENTIONS:
Procedure: High Flow oxygen — 10 minute shigh flow oxygen
  Arms: High Flow oxygen
Procedure: Room Air — Room air breathing
  Arms: Room Air

SUMMARY:
Coronary artery disease (CAD) is a condition which refers to the narrowing of the small blood vessels that supplies blood and oxygen to the heart. It is a common cause of chest-pain related symptoms and as a result of a 'heart attack'. In most cases, to assess the severity of the disease is to use coronary angiography, which is a medical imaging technique that uses contrast (a dye) and x-ray to show the blood-flow supply of the coronary arteries.

The optimal treatment for patients with symptomatic coronary disease is aggressive medical therapy. Current guidelines recommend patients with symptomatic CAD and severe disease on angiography undergo revascularisation therapy, which aims to restore blood flow to blocked arteries. This can be done by either percutaneous coronary intervention (feeding a small balloon or other device on a thin tube through blood vessels to the point of blockage and then inflate the balloon to open the artery), or coronary artery bypass grafting (open-heart surgery)2.

For many symptomatic patients who have only moderate disease on angiography, further functional testing is required to assess the extent of the blockage. This can be achieved by placing a pressure wire to the artery of interest, to determine the likelihood that the blockage impedes oxygen delivery to the heart muscle, known as the Fractional Flow Reserve (FFR)3. FFR is commonly performed at the Alfred hospital in the assessment of such patients. During an FFR procedure, further information regarding the health of the small arteries of the heart can be obtained with the calculation of the index of micro-vascular resistance (IMR),

Giving oxygen to patients with CAD is a common clinical practice, especially to all patients in the catheterisation laboratory whose had a 'heart attack' and often administered concurrently with light sedation during elective procedures.

Recently, however, the safety of routine supplemental oxygen in patients with CAD has been questioned5. A research study analysed the outcomes of three small randomised studies on oxygen in patients who experienced a 'heart attack', while suggestive of harm, the findings of the study remain inconclusive.

There may also be deleterious effects of supplemental oxygen, on more stable patients with CAD, who are not experiencing a 'heart attack'. Supplemental oxygen administered in the catheterisation laboratory to patients with stable CAD, has been shown to significantly reduce coronary artery blood flow and increase its resistance6-8. It has also been shown to reduce cardiac output and effect the relaxation phase of the heart cycle. Based on this data it is hypothesised that supplemental oxygen may affect FFR in patients with moderate CAD. The investigators therefore propose to undertake a study of the effects of supplemental oxygen on FFR in patients with moderate CAD.

The patients enrolled into the study will be scheduled for an elective normal contrast diagnostic or interventional procedure as part of their clinically-indicated care. Once a moderate blockage of the artery has been identified, FFR and IMR will be measured. During the first phase of the FFR study, the patient will breathe room air and have a blood test to measure their oxygen level (blood gas). There is a 3 minute washout period, followed by the second phase, whereby the patient will be given 100% oxygen for 10 minutes and have another blood gas measured.

The study will be conducted at Alfred Hospital with a total enrollment of 18 subjects. The estimated time to complete enrollment is 6-10 months.

Data collected on each patient will include demographics, medical history, vital signs (heart rate, blood pressure, height, and weight), usage of cardiovascular medications, pathology results and procedural records. Any adverse events or serious adverse events related to the study procedure will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age, AND
* Undergoing elective coronary angiography
* Evidence of moderate (40%-79%) stenosis, requiring further routine assessment with FFR.

Exclusion Criteria:

* Acute coronary syndrome
* Hypoxia with oxygen saturation measured on pulse oximeter < 94% with the patient breathing air
* Altered conscious state
* Evidence of left ventricular failure or cardiogenic shock
* Unable to perform consent prior to procedure
* Known hypersensitivity to adenosine
* Sick sinus syndrome, second or third degree atrioventricular (A-V) block (except in patients with a functioning artificial pacemaker).
* Chronic Obstructive lung disease COPD or asthma
* Long QT syndrome
* Severe hypotension
* Concomitant use of dipyridamole

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Fractional flow reserve | Duration of inpatient stay 2-3 days

SECONDARY OUTCOMES:
index of micro-vascular resistance | Duration of inpatient stay 2-3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia